CLINICAL TRIAL: NCT05656599
Title: Immune Reconstitution to Cytomegalovirus After Allogeneic Hematopoietic Stem Cell Transplantation: Impact of Clinical Factors and Therapy Strategies
Brief Title: Immune Reconstitution to CMV After HSCT: Impact of Clinical Factors and Therapy Strategies
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Chairman of the department, Peking University People's Hospital
Other Study IDs: 2021PHB423-001
Record Dates: First submitted 2022-11-25; First posted 2022-12-19 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: CMV Infection; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Letermovir Group: HSCT recipients who received letermovir prophylaxis
  Interventions: Drug: Letermovir
- Preemptive therapy Group: HSCT recipients who received PCR-guided preemptive therapy

INTERVENTIONS:
Drug: Letermovir — Patients received letermovir as prophylaxis or received preemptive therapy for CMV depends on clinical needs and patients' wishes
  Groups: Letermovir Group

SUMMARY:
Cytomegalovirus (CMV) remains a significant cause of morbidity and mortality after hematopoietic stem cell transplantation (HSCT). The course and outcome of CMV infection are different clinically, and the mechanism of CMV infection after transplantation has not been clarified. Reconstitution of cellular immunity after HSCT is a critical determinant of the control of CMV infection.

Investigators will dynamically monitor the CMV-specific cellular immune reconstitution after HSCT，and analyze the clinical factors and therapy strategies affecting recovery of CMV-specific immunity during 1 year after HSCT.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) remains a significant cause of morbidity and mortality after hematopoietic stem cell transplantation (HSCT). The course and outcome of CMV infection are different clinically, and the mechanism of CMV infection after transplantation has not been clarified. Reconstitution of cellular immunity after HSCT is a critical determinant of the control of CMV infection.

Investigators will collect peripheral blood at 1 month, 2 month, 3 month, and 6 month after HSCT from the participated patients, and dynamically monitor the CMV-specific T and NK cellular immune reconstitution.

Investigators will also analyze the clinical factors and therapy strategies affecting recovery of CMV-specific immunity during 1 year after HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Be receiving a first allogeneic HSCT.
* Is male or female, from 14 years to any years of age inclusive.
* The participant (or legally acceptable representative) agree for cellular immune investigation and has provided documented informed consent/assent for the study.

Exclusion Criteria:

* Received a previous allogeneic HSCT (Note: Receipt of a previous autologous HSCT is acceptable).
* Has a history of CMV end-organ disease within 6 months prior to allocation.
* Has severe organ (hepatic , renal, cardical) insufficiency within 5 days prior to allocation.
* Any rapidly-progressing disease or immediately life-threatening illness.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients who received allogeneic HSCT.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically significant CMV infection (CSI) | 6 months after HSCT
  Clinically significant CMV infection (CSI) is defined as the administration of antiviral therapy as preemptive therapy for CMV DNAemia or treatment for CMV disease.
Incidence of refractory CMV infection and CMV disease | 6 months after HSCT
  Refractory CMV infection is defined as a persistent viral load (CMV viral load at the same level or higher than the peak viral load within 1 week but <1 log10 increase in CMV DNA titers done in the same laboratory and with the same assay) after at least 2 weeks of appropriately dosed antiviral therapy.
Numbers of immune cells in peripheral blood | 6 months after HSCT
  PBMCs from HSCT recipients were collected at 1 month, 2 month, 3 month, and 6 month after HSCT, and tested for NK cells, T cells, CMV-specific T cells and their subsets.

SECONDARY OUTCOMES:
Treatment-ralated mortality | Through study completion, an average of 1 year
  Treatment-ralated mortality
Overall survival | Through study completion, an average of 1 year
  Overall survival
Incidence of other viral infection and viral-associated disease | 6 months after HSCT
  Other viral infection and viral-associated diseases including EBV, ADV, HHV-6, BKV and HSV

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality
  - People's Hospital of Peking University, Beijing